CLINICAL TRIAL: NCT05360927
Title: A Randomized, Double-blind,Placebo-controlled,Single-Ascending Dose Phase Ⅰ Study to Evaluate the Safety,Tolerability,and Pharmacokinetics of BDB-001 Injection in Healthy Subjects
Brief Title: Safety and Tolerability of BDB-001 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Collaborators: Beijing Defengrei Biotechnology Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STS-BDB001-01
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — BDB001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 0.3mg/kg (Experimental): All participants (fasted) received either 0.3 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 1mg/kg (Experimental): All participants (fasted) received either 1 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 3mg/kg (Experimental): All participants (fasted) received either 3 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 8mg/kg (Experimental): All participants (fasted) received either 8 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 16mg/kg (Experimental): All participants (fasted) received either 16 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo
- Cohort 20mg/kg (Experimental): All participants (fasted) received either 20 mg/kg of BDB-001 as a single dose or dose-matched placebo.
  Interventions: Drug: BDB-001 injection; Drug: Placebo

INTERVENTIONS:
Drug: BDB-001 injection — Intravenous injection
Drug: Placebo — Intravenous injection

SUMMARY:
A clinical study to evaluate the safety,tolerability,PK and PD characteristics of BDB-001 Injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 but ≤ 65, male and female;
* Medical histories, physical examinations, laboratory examinations and study-related examinations and tests of the subjects，the Investigator judges that they are healthy;
* Body weight: 50- 80 kg, inclusive; Body mass index: 18.0 -26.0 kg/m2, inclusive;
* Vital signs: Blood pressure (90 mmHg≤ systolic ≤140 mmHg, 50 mmHg≤ diastolic ≤90 mmHg), heart rate (50≤ heart rate ≤100 beats/min), body temperature < 37°C;
* Subjects (including their partners) agree to take highly effective contraceptive measures during the study, and they have no birth plan or sperm donation plan within 6 months after the end of the study;
* Subjects are aware of the risks of the study, and voluntarily participate in the clinical study and sign an informed consent form (ICF).

Exclusion Criteria:

* History of cardiovascular, respiratory, kidney, liver, metabolism, endocrine, gastrointestinal, blood, nerve, skin and mental illness, cancer or other major disease that in the judgment of the Investigator might put the subject as risk on this study;
* Past history of tuberculosis, history of contact with active tuberculosis, TB-SPOT test results exceeding the upper limit of 2 times or more, and recent infectious diseases;
* During the screening and baseline period, the white blood cell count and C-reactive protein test results are abnormal and have clinical significance, hemoglobin: male <120g/L or female <110g/L;
* Electrocardiogram (ECG) abnormalities and have clinical significance;
* Subjects who have an autoimmune disease or an immune deficiency disease, or a family history of an autoimmune disease or an immune deficiency disease;
* Subjects with clinically obvious allergic diseases;
* Positive screening test results for human immunodeficiency virus (HIV-1/HIV-2) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab), treponema pallidum antibody;
* Participate in any drug or vaccine clinical trial as a subject within 3 months before screening or prepare to be vaccinated during the study period to 2 months after the end of the study;
* Have received any monoclonal antibody or biological agent treatment within the previous 3 months;
* Have taken drugs that may affect immune function within 6 months before screening or have taken prescription/over-the-counter drugs within the previous 14 days;
* Subjects who have donated either more than approximately 500 mL of blood within 3 months prior to screening or any plasma within 4 weeks prior to screening; Subjects who donated blood (>400 ml) within 3 months prior to screening, or plasma exchange within 4 weeks prior to screening;
* Drink more than 5 cups of coffee, tea or cola per day (150ml and above per cup);
* Subjects who test positive for alcohol or drugs during the screening;
* Subjects who smoke or smoke test results are positive;
* Subjects with poor compliance;
* Pregnant or lactating women;
* The investigator believes that there are any subjects who are not suitable to participate in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram Abnormalities, Clinically Significant Vital Signs Abnormalities And Clinically Significant Physical Examination Abnormalities | Up to 50 days
Maximum plasma concentration (Cmax) | Up to 1200 hours postdose
Area under the plasma concentration-time curve from time 0 to infinity (AUC0inf) | Up to 1200 hours postdose
Area under the plasma concentration-time curve from time 0 to 1200hr(AUC00-1200hr) | Up to 1200 hours postdose
Time of maximum concentration (Tmax) | Up to 1200 hours postdose
Elimination half-life (t1/2) | Up to 1200 hours postdose
Clearance (CL) | Up to 1200 hours postdose
Apparent volume of distribution (Vz) | Up to 1200 hours postdose
Mean residence time (MRT) | Up to 1200 hours postdose

SECONDARY OUTCOMES:
Number of participants developing anti-BDB-001 antibodies | Up to 50 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No